CLINICAL TRIAL: NCT00854633
Title: Phase 1/2 Study of Talactoferrin Oral Solution for Nosocomial Infection in Preterm Infants
Brief Title: Study of Talactoferrin Oral Solution for Nosocomial Infection in Preterm Infants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Agennix (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LF-0901; 1R44HD057744-01A1 (NIH)
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Nosocomial Infections
Keywords: Pre-term infants; Pre-term infants 750 to 1500 grams
MeSH Terms: conditions — Cross Infection | interventions — talactoferrin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Talactoferrin
  Interventions: Drug: Talactoferrin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Talactoferrin — Enteral, 150 mg/kg twice per day
  Other Names: talactoferrin alfa; TLF; recombinant human lactoferrin; rhLF
  Arms: 1
Drug: Placebo — Oral, twice per day
  Arms: 2

SUMMARY:
This study will evaluate the safety, toxicity and efficacy of talactoferrin in reducing the incidence of all nosocomial infections in prematurely-born infants.

ELIGIBILITY:
Inclusion Criteria:

* Birth weights ranging from 750 to 1500 grams
* Entry before 24 hours of age
* Informed-consent form signed by parent(s) or legal guardian
* Able to take liquid medication by mouth or feeding tube

Exclusion Criteria

* A major birth defect or malformation syndrome
* Chromosomal or inherited disorder
* Proven presence of an immunodeficiency
* Antenatal exposure to illicit substances
* Birth asphyxia
* HIV or other congenital viral, bacterial, or fungal infection
* Lack of parental consent or refusal of attending neonatologist to allow participation
* Discretion of the investigator
* The legal representative of the infant or the patient's primary physician are not committed to providing full, aggressive life support

Ages: 1 Minute to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in incidence of Late-Onset Infection defined by positive cultures and elevated C-reactive protein (CRP) | 1-3 months

SECONDARY OUTCOMES:
"NEC Scares", the "Neonatal Sepsis Syndrome" | 1-3 months
Length of stay: The number of days of hospitalization from the date of birth until the day of discharge from the NICU | 1-3 months
Mortality during hospitalization | 1-3 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Kosair Children's Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Missouri Health Care, Columbia Regional Hospital, Columbia, Missouri

REFERENCES:
- [Derived] Sherman MP, Adamkin DH, Niklas V, Radmacher P, Sherman J, Wertheimer F, Petrak K. Randomized Controlled Trial of Talactoferrin Oral Solution in Preterm Infants. J Pediatr. 2016 Aug;175:68-73.e3. doi: 10.1016/j.jpeds.2016.04.084. Epub 2016 May 31. PMID 27260839
- [Derived] Sherman MP, Sherman J, Arcinue R, Niklas V. Randomized Control Trial of Human Recombinant Lactoferrin: A Substudy Reveals Effects on the Fecal Microbiome of Very Low Birth Weight Infants. J Pediatr. 2016 Jun;173 Suppl:S37-42. doi: 10.1016/j.jpeds.2016.02.074. PMID 27234409